CLINICAL TRIAL: NCT03014089
Title: A Phase 1, Randomized, Placebo-Controlled, Dose-Ranging Study to Evaluate the Safety and Immunogenicity of mRNA 1325 Zika Vaccine in Healthy Adults in a Non-endemic Zika Region
Brief Title: Safety, Tolerability, and Immunogenicity of mRNA-1325 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: mRNA-1325-P101; HHSO100201600029C (Other Grant/Funding Number: Biomedical Advanced Research & Development Authority (BARDA))
Record Dates: First submitted 2017-01-05; First posted 2017-01-09 (Estimated); Results first posted 2024-06-17 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-07

CONDITIONS: Zika Virus
Keywords: mRNA-1325; Zika vaccine
MeSH Terms: conditions — Zika Virus Infection

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- mRNA-1325 (Experimental)
  Interventions: Biological: mRNA-1325
- Placebo (Placebo Comparator): 0.9% sodium chloride
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: mRNA-1325 — Escalating dose levels
  Arms: mRNA-1325
Other: Placebo
  Arms: Placebo

SUMMARY:
The clinical study will assess the safety, tolerability, and immunogenicity of mRNA-1325 in healthy adult subjects.

ELIGIBILITY:
Inclusion

* 18 to 49 years of age
* Body mass index between 18 and 35 kg/m2
* In good health as determined by medical history
* Female subjects must be non pregnant and non lactating and meet one of the following criteria: a) post menopausal b) surgically sterile
* Women of childbearing potential must agree to be heterosexually inactive or agree to consistently use any of the following methods of contraception from at least 21 days prior to enrollment and through 3 months after the final vaccination
* Male subjects must use an acceptable method of birth control throughout the entire study and agree to refrain from donation of sperm from the time of first vaccination until 3 months following the last vaccination
* Agrees to comply with the study procedures and provides written informed consent
* Has access to a consistent and reliable means of telephone contact and agrees to stay in contact with the study site for the duration of the study, to provide updated contact information as necessary, and has no current plans to move from the study area for the duration of the study

Exclusion

* Any ongoing, symptomatic acute or chronic illness requiring medical or surgical care
* A history of active cancer (malignancy) in the last 10 years
* Female of childbearing potential and has a positive pregnancy test at screening or on the day of vaccination
* Administration of an investigational product within 60 days, or 5 half-lives, whichever is longer
* Administration of any live attenuated vaccines within 4 weeks before enrollment or inactive vaccines within 2 weeks before enrollment, or plans to receive any vaccine during the active vaccination period
* Prior administration of a vaccine for Zika or dengue vaccine, a history of confirmed Zika or dengue infection, or has lived in or visited any Zika-endemic area greater than 4 weeks in duration
* Prior administration of investigational agent using formulations similar to mRNA-1325
* A history of hypersensitivity or serious reactions to previous vaccinations
* Any known or suspected autoimmune disease or immunosuppressive condition, acquired or congenital, as determined by medical history and/or physical examination
* A history of inflammatory arthritis
* Any neurologic disorder
* A history of febrile disease with arthritis or arthralgia within 2 weeks of dose administration.
* Prior administration of immunoglobulins and/or any blood products within the 3 months preceding the administration of the study drug or plans to receive such products at any time during the study
* Any chronic administration of an immunosuppressant or other immune modifying drug
* Any acute illness at the time of enrollment
* Any significant disorder of coagulation requiring ongoing or intermittent treatment
* A history of idiopathic urticaria
* A history of alcohol abuse or drug addiction
* A positive test result for drugs of abuse
* The subject has any abnormality or permanent body art (eg, tattoo) that, in the opinion of the investigator, would obstruct the ability to observe local reactions at the injection site
* Any condition that, in the opinion of the investigator, would pose a health risk to the subject if enrolled or could interfere with evaluation of the study drug or interpretation of study results
* A positive test result for hepatitis B surface antigen, hepatitis C virus antibody, or human immunodeficiency virus types 1 or 2 antibodies
* Donation of blood or blood products > 450 mL within 30 days of dosing.
* Abnormal vital signs or screening safety laboratory test results including liver enzyme tests
* Is an employee or first degree relative of the Sponsor, CRO, or study site personnel

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2016-12-21 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - San Diego, California
  - Melbourne, Florida
  - Peoria, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Essink B, Chu L, Seger W, Barranco E, Le Cam N, Bennett H, Faughnan V, Pajon R, Paila YD, Bollman B, Wang S, Dooley J, Kalidindi S, Leav B. The safety and immunogenicity of two Zika virus mRNA vaccine candidates in healthy flavivirus baseline seropositive and seronegative adults: the results of two randomised, placebo-controlled, dose-ranging, phase 1 clinical trials. Lancet Infect Dis. 2023 May;23(5):621-633. doi: 10.1016/S1473-3099(22)00764-2. Epub 2023 Jan 19. PMID 36682364

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a 2-part study. Part A was conducted for 28 days following the second vaccination. Once the participants completed the final visit in Part A, they were entered into Part B. Part B was conducted for 12 months following the second vaccination in Part A.
Groups:
- mRNA-1325 10 mcg: Participants received mRNA-1325 10 micrograms (mcg) intramuscular (IM) injection on Days 1 and 29.
- mRNA-1325 25 mcg: Participants received mRNA-1325 25 mcg as an IM injection on Days 1 and 29.
- mRNA-1325 100 mcg: Participants received mRNA-1325 100 mcg as an IM injection on Days 1 and 29.
- Placebo: Participants received placebo matched to mRNA-1325 as an IM injection on Days 1 and 29.
Period: Overall Study
Arm/Group | mRNA-1325 10 mcg | mRNA-1325 25 mcg | mRNA-1325 100 mcg | Placebo
Started | 25 | 24 | 25 | 16
Received Injection 1 | 25 | 24 | 25 | 16
Received Injection 2 | 25 | 24 | 24 | 16
Completed | 23 | 23 | 23 | 15
Not Completed | 2 | 1 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Safety set included all participants in Randomized Set who received at least 1 dose of study drug (mRNA-1325 or placebo).
Groups:
- mRNA-1325 10 mcg: Participants received mRNA-1325 10 mcg IM injection on Days 1 and 29.
- Total: Total of all reporting groups
Arm/Group | mRNA-1325 10 mcg | mRNA-1325 25 mcg | mRNA-1325 100 mcg | Placebo | Total
Number analyzed (Participants) | 25 | 24 | 25 | 16 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.9 (8.57) | 34.4 (9.42) | 35.3 (8.59) | 38.9 (8.69) | 35.3 (8.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 14 | 13 | 10 | 53
  Male | 9 | 10 | 12 | 6 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 5 | 1 | 2 | 15
  Not Hispanic or Latino | 17 | 19 | 24 | 14 | 74
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 1 | 0 | 3
  White | 23 | 22 | 24 | 15 | 84
  More than one race | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Part A: Number of Participants With Solicited Adverse Events- Vaccination 1
Description: Solicited adverse reactions (ARs) (local and systemic) were collected in the electronic diary (eDiary). Local ARs included: injection site pain, injection site erythema, and injection site induration/swelling. Systemic ARs included: body temperature (oral), generalized myalgia (muscle ache or pain), generalized arthralgia (joint ache or pain), headache, fatigue/malaise (unusual tiredness), nausea/vomiting, chills, and rash. Data for this outcome measure is reported up to 7 days after the first study vaccination only. A summary of all serious AEs (SAEs) and nonserious AEs ("Other"), regardless of causality, is in Reported "Adverse Events" section.
Time Frame: Up to 7 days post-vaccination 1 (up to 8 days)
Population: The Safety set included all participants in Randomized Set who received at least 1 dose of study drug (mRNA-1325 or placebo) and provided vaccination 1 safety data.
Measure: Count of Participants; unit: Participants
Arm/Group | mRNA-1325 10 mcg | mRNA-1325 25 mcg | mRNA-1325 100 mcg | Placebo
Number analyzed (Participants) | 25 | 24 | 25 | 16
Participants
  Local Event- Pain | 17 | 20 | 24 | 0
  Local Event- Tenderness | 21 | 20 | 23 | 3
  Local Event- Swelling | 0 | 1 | 1 | 0
  Local Event- Redness | 0 | 0 | 1 | 0
  Systemic Event- Fever | 0 | 0 | 2 | 1
  Systemic Event- Vomiting | 3 | 0 | 2 | 0
  Systemic Event- Diarrhea | 2 | 0 | 0 | 0
  Systemic Event- Headache | 11 | 4 | 10 | 3
  Systemic Event- Fatigue | 7 | 4 | 4 | 2
  Systemic Event- Generalized Myalgia | 8 | 9 | 11 | 0
  Systemic Event- Generalized Arthralgia | 3 | 3 | 5 | 0

2. Primary Outcome: Part A: Number of Participants With Solicited Adverse Events: Vaccination 2
Description: Solicited adverse reactions (ARs) (local and systemic) were collected in the electronic diary (eDiary). Local ARs included: injection site pain, injection site erythema, and injection site induration/swelling. Systemic ARs included: body temperature (oral), generalized myalgia (muscle ache or pain), generalized arthralgia (joint ache or pain), headache, fatigue/malaise (unusual tiredness), nausea/vomiting, chills, and rash. Data for this outcome measure is reported up to 7 days after the second study vaccination only. A summary of all serious AEs (SAEs) and all nonserious AEs ("Other"), regardless of causality, is in Reported "Adverse Events" section.
Time Frame: Up to 7 days post-vaccination 2 (Day 29 to Day 36)
Population: The Safety set included all participants in Randomized Set who received at least 1 dose of study drug (mRNA-1325 or placebo) and provided post vaccination 2 safety data.
Measure: Count of Participants; unit: Participants
Arm/Group | mRNA-1325 10 mcg | mRNA-1325 25 mcg | mRNA-1325 100 mcg | Placebo
Number analyzed (Participants) | 25 | 24 | 24 | 16
Participants
  Local Event- Pain | 19 | 19 | 19 | 1
  Local Event- Tenderness | 22 | 19 | 20 | 0
  Local Event- Swelling | 0 | 0 | 1 | 0
  Local Event- Redness | 1 | 0 | 2 | 0
  Systemic Event- Fever | 1 | 2 | 7 | 0
  Systemic Event- Vomiting | 4 | 4 | 7 | 0
  Systemic Event- Diarrhea | 2 | 0 | 1 | 0
  Systemic Event- Headache | 9 | 11 | 10 | 2
  Systemic Event- Fatigue | 11 | 12 | 11 | 0
  Systemic Event- Generalized Myalgia | 13 | 10 | 12 | 0
  Systemic Event- Generalized Arthralgia | 6 | 7 | 6 | 0

3. Primary Outcome: Part A: Number of Participants With Unsolicited Adverse Events
Description: An unsolicited AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. The treatment-emergent AEs are defined as any event not present before exposure to study drug or any event already present that worsened in intensity or frequency after exposure. A summary of all SAEs and all nonserious AEs ("Other") reported up to the end of the study, regardless of causality, is located in the Reported "Adverse Events" section.
Time Frame: Up to Day 392 (all AEs considered an SAE were collected till end of study [Day 392]; the Other AEs [non-SAE] were collected up to Day 57)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | mRNA-1325 10 mcg | mRNA-1325 25 mcg | mRNA-1325 100 mcg | Placebo
Number analyzed (Participants) | 25 | 24 | 25 | 16
Participants | 14 | 9 | 14 | 6

4. Primary Outcome: Part A: Number of Participants With Medically-Attended Adverse Events (MAAEs)
Description: An MAAE is an AE that leads to an unscheduled visit to an healthcare practitioner. A summary of all SAEs and all nonserious AEs ("Other"), regardless of causality, is located in the Reported "Adverse Events" section.
Time Frame: Up to 1 year post-vaccination (Day 392)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | mRNA-1325 10 mcg | mRNA-1325 25 mcg | mRNA-1325 100 mcg | Placebo
Number analyzed (Participants) | 25 | 24 | 25 | 16
Participants | 5 | 3 | 3 | 1

5. Primary Outcome: Part B: Number of Participants With Adverse Events of Special Interest (AESIs) and Serious Adverse Events (SAEs)
Description: An SAE was defined as any AE that resulted in death, is life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions was a congenital anomaly/birth defect, or was an important medical event. AESIs included potentially immune-mediated medical conditions (autoimmune or autoinflammatory diseases) that may have the theoretical potential for association with novel vaccines. A summary of all SAEs and all nonserious AEs ("Other"), regardless of causality, is located in the Reported "Adverse Events" section.
Time Frame: Up to 1 year post-vaccination (Day 392)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | mRNA-1325 10 mcg | mRNA-1325 25 mcg | mRNA-1325 100 mcg | Placebo
Number analyzed (Participants) | 25 | 24 | 25 | 16
Participants
  AESI | 0 | 0 | 0 | 0
  SAE | 1 | 0 | 0 | 0

6. Secondary Outcome: Part A: Geometric Mean Titer of Neutralizing Serum Antibody (PRNT50) to Zika Virus
Description: GMT 95% CI is calculated based on the t-distribution of the log-transformed values, then back transformed to the original scale for presentation.
Time Frame: Baseline, 28 days post each vaccination (Days 29 and 57)
Population: The per-protocol set included all participants in the randomized set who did not have a major protocol violation, received the full dose of the assigned investigational product within the acceptable vaccination window, had blood collection within accepted visit windows, and had a pre-vaccination and at least 1 serum sample from the post-vaccination immunogenicity testing period available for testing. Here, number analyzed signifies those participants who were evaluable at specified time points.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | mRNA-1325 10 mcg | mRNA-1325 25 mcg | mRNA-1325 100 mcg | Placebo
Number analyzed (Participants) | 25 | 24 | 25 | 16
Titer
  Baseline: number analyzed (Participants) | 24 | 24 | 25 | 16
  Baseline | 5.4 [4.6 to 6.4] | 5.0 [NA to NA] — All values were equal to 5.0, therefore CI (upper and lower limit) could not be calculated. | 5.0 [NA to NA] — All values were equal to 5.0, therefore CI (upper and lower limit) could not be calculated. | 5.0 [NA to NA] — All values were equal to 5.0, therefore CI (upper and lower limit) could not be calculated.
  Day 29: number analyzed (Participants) | 24 | 22 | 23 | 15
  Day 29 | 5.8 [4.2 to 8.0] | 5.6 [4.8 to 6.6] | 5.2 [4.8 to 5.7] | 5.0 [NA to NA] — All values were equal to 5.0, therefore CI (upper and lower limit) could not be calculated.
  Day 57: number analyzed (Participants) | 24 | 24 | 22 | 16
  Day 57 | 10.3 [5.9 to 18.2] | 6.6 [4.8 to 9.0] | 7.7 [5.2 to 11.4] | 5.0 [NA to NA] — All values were equal to 5.0, therefore CI (upper and lower limit) could not be calculated.

ADVERSE EVENTS:
Time Frame: Baseline up to Day 392
Description: The Safety set included all participants in Randomized Set who received at least 1 dose of study drug (mRNA-1325 or placebo). Adverse Events reported in the Adverse Events section below include unsolicited AEs and solicited ARs. All AEs considered an SAE were collected till end of study (Day 392). The Other AEs (non-SAE) were collected up to Day 57. All cause mortality includes the deaths that were due to "AEs leading to death".
Groups:
- mRNA-1325 25 mcg: Participants received placebo matched to mRNA-1325 as an IM injection on Days 1 and 29.
- mRNA-1325 100 mcg: Participants received mRNA-1325 25 mcg as an IM injection on Days 1 and 29.
- Placebo: Participants received mRNA-1325 100 mcg as an IM injection on Days 1 and 29.
Arm/Group | mRNA-1325 10 mcg | mRNA-1325 25 mcg | mRNA-1325 100 mcg | Placebo
All-Cause Mortality (participants affected / at risk) | 1/25 | 0/24 | 0/25 | 0/16
Serious Adverse Events (participants affected / at risk) | 1/25 | 0/24 | 0/25 | 0/16
Other Adverse Events (participants affected / at risk) | 24/25 | 23/24 | 25/25 | 12/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | mRNA-1325 10 mcg (N=25) | mRNA-1325 25 mcg (N=24) | mRNA-1325 100 mcg (N=25) | Placebo (N=16)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | mRNA-1325 10 mcg (N=25) | mRNA-1325 25 mcg (N=24) | mRNA-1325 100 mcg (N=25) | Placebo (N=16)
Pharyngitis streptococcal (Infections and infestations) | 0 | 2 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0
Ear infection (Infections and infestations) | 0 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 1
Headache (Nervous system disorders) | 14 | 11 | 14 | 6
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 7 | 4 | 7 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 16 | 14 | 15 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 8 | 8 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Injection site lymphadenopathy (General disorders) | 23 | 20 | 25 | 3
Injection site pain (General disorders) | 21 | 22 | 25 | 1
Fatigue (General disorders) | 14 | 13 | 13 | 2
Pyrexia (General disorders) | 1 | 2 | 7 | 1
Injection site erythema (General disorders) | 1 | 0 | 2 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 1 | 0
Injection site induration (General disorders) | 0 | 1 | 1 | 0
Influenza like illness (General disorders) | 1 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 1 | 0
Lipase increased (Investigations) | 0 | 1 | 4 | 1
Haemoglobin decreased (Investigations) | 1 | 0 | 0 | 0
Red blood cells urine positive (Investigations) | 0 | 0 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Animal bite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Corneal abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (3):
  • Study Protocol (2018-08-13): https://cdn.clinicaltrials.gov/large-docs/89/NCT03014089/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-15): https://cdn.clinicaltrials.gov/large-docs/89/NCT03014089/SAP_001.pdf
  • Informed Consent Form (2017-06-13): https://cdn.clinicaltrials.gov/large-docs/89/NCT03014089/ICF_002.pdf